CLINICAL TRIAL: NCT00853151
Title: A Proof of Concept Study to Evaluate the Coadministration of TT223 Given Daily and LY2428757 Given Once-Weekly for Four Weeks in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Test the Combination of Two Different Kinds of Medications for the Treatment of Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12758; I3H-MC-GAFA(b) (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LY2428757 plus TT223 3 milligrams (mg) (Experimental): Weekly LY2428757 plus 3 milligrams (mg) daily TT223
  Interventions: Drug: LY2428757; Drug: TT223
- LY2428757 plus TT223 2mg (Experimental): Weekly LY2428757 plus 2 mg daily TT223
  Interventions: Drug: LY2428757; Drug: TT223
- LY2428757 plus placebo (Experimental): Weekly LY2428757 plus daily TT223 placebo
  Interventions: Drug: LY2428757; Drug: Placebo for TT223
- Placebo plus Placebo (Placebo Comparator): Weekly LY2428757 placebo plus daily TT223 placebo
  Interventions: Drug: Placebo for LY2428757; Drug: Placebo for TT223

INTERVENTIONS:
Drug: LY2428757 — 14 mg subcutaneous injection 1 time a week for 5 weeks
  Arms: LY2428757 plus TT223 2mg; LY2428757 plus TT223 3 milligrams (mg); LY2428757 plus placebo
Drug: TT223 — subcutaneous injection once a day for 4 weeks
  Arms: LY2428757 plus TT223 2mg; LY2428757 plus TT223 3 milligrams (mg)
Drug: Placebo for LY2428757 — subcutaneous injection 1 time a week for 5 weeks
  Arms: Placebo plus Placebo
Drug: Placebo for TT223 — subcutaneous injection once a day for 4 weeks
  Arms: LY2428757 plus placebo; Placebo plus Placebo

SUMMARY:
Test the safety, tolerability and improvement of blood sugar control with combination therapy in individuals with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Have type 2 diabetes mellitus (T2DM) for at least 6 months
* Currently treated with diet and exercise alone or in combination with stable metformin
* Glycosylated hemoglobin (HbA1c) 7.0% to 10.0%
* Ages 18 to 70 years
* Women not of childbearing potential
* Body mass index (BMI) between 25 and 40 kilograms per meters squared (kg/m^2), and stable weight in the 3 months prior to screening.

Exclusion Criteria:

* Use of diabetes medicine other than metformin in past 3 months
* Gastrointestinal disease or surgery or drugs that significantly impacts gastric filling, emptying or motility; ongoing cholelithiasis or cholecystitis.
* Chronic, daily proton pump inhibitors (PPIs) and histamine (H2) antagonists.
* Severe hypoglycemia or hyperglycemia
* Advanced microvascular diabetes complications
* Medications to promote weight loss.
* Breastfeeding women
* Cardiac autonomic neuropathy
* In the past 6 months have cardiac disease with functional status that is Class II-IV or a history of myocardial infarction, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, transient ischemic attack, cerebrovascular accident (stroke), or decompensated congestive heart failure.
* History of a supraventricular or ventricular tachycardia, pacemaker implantation, or other cardiac arrhythmia: Poorly controlled hypertension, malignant hypertension, renal artery stenosis, and/or evidence of labile blood pressure including symptomatic postural hypotension.
* Electrocardiograms (ECG) abnormality or medication that impairs the ability to measure QT interval (QT), or correct the QT interval (QT) for rate.
* QT interval Bazett corrected (QTcB) >450 milliseconds (msec) or PR interval (PR) >220 milliseconds (msec)
* Personal or family history of long QT interval (QT) syndrome, sudden death, or unexplained syncope
* Clinical signs or symptoms of liver disease, acute or chronic hepatitis, or alanine transaminase levels > 2.5 times the upper limit of the reference range
* Hypertriglyceridemia > 400 mg/deciliter (dL)
* Inadequately treated hypothyroidism or hyperthyroidism
* Peptic ulcer disease and/or gastrointestinal bleeding/perforation.
* Known pentagastrin hypersensitivity
* Impaired renal function
* Transplanted organ.
* Active, uncontrolled endocrine or autoimmune abnormality
* > 2 weeks systemic glucocorticoid therapy
* Ongoing courses of non-steroidal anti-inflammatory drugs (NSAIDs), except for aspirin 81-325 milligrams (mg)
* Diagnosed malignancy or in remission for less than 5 years.
* Prior acute or chronic pancreatitis or elevated serum lipase or amylase
* Current central nervous system stimulant
* Other conditions that preclude the participant from participating, following or completing the protocol.
* Chronic infection
* Personnel affiliated with the study and their immediate families.
* Within 30 days of the initial dose of study drug, have participated in an interventional medical, surgical, or pharmaceutical study in which a medical or surgical treatment was given.
* Have previously completed or withdrawn from this study after providing informed consent.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- United States (26):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Artesia, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norwalk, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yukon, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taylors, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingsport, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midvale, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Virginia Beach, Virginia
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Reporting on 131 participants who received either TT223 or its placebo and reflects data from treatment and follow-up. 151 enrolled in run-in. 16/130 randomized to LY2428757 run-in did not get treatment assignment. 3/21 assigned to placebo run-in did not enter treatment phase. 1 was given treatment assignment but never received TT223 or placebo.
Groups:
- LY2428757 Plus TT223 3mg: Weekly LY2428757 14 mg subcutaneous injection for 5 weeks plus TT223 3 mg subcutaneous injection daily for 4 weeks
- LY2428757 Plus TT223 2mg: Weekly LY2428757 14 mg subcutaneous injection for 5 weeks plus TT223 2 mg subcutaneous injection daily for 4 weeks
- LY2428757 Plus TT223 Placebo: Weekly LY2428757 14 mg subcutaneous injection for 5 weeks plus TT223 placebo subcutaneous injection daily for 4 weeks
- LY Placebo Plus TT223 Placebo: Weekly LY2428757 placebo subcutaneous injection for 5 weeks plus TT223 placebo subcutaneous injection daily for 4 weeks
Period: Overall Study
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Started | 38 | 37 | 38 | 18
Completed | 28 | 24 | 30 | 15
Not Completed | 10 | 13 | 8 | 3
Not completed — Adverse Event | 1 | 4 | 2 | 0
Not completed — Inclusion/Exclusion Criteria Not Met | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 3 | 0
Not completed — Death | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 4 | 2 | 1
Not completed — Physician Decision | 0 | 2 | 1 | 0
Not completed — Sponsor Decision | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo | Total
Number analyzed (Participants) | 38 | 37 | 38 | 18 | 131
Age Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.69) | 52.4 (10.12) | 52.9 (8.99) | 55.4 (7.90) | 53.3 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 16 | 5 | 55
  Male | 21 | 20 | 22 | 13 | 76
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan Native | 0 | 1 | 0 | 1 | 2
  Asian | 2 | 0 | 1 | 1 | 4
  Black or African American | 4 | 3 | 4 | 3 | 14
  White | 32 | 31 | 33 | 12 | 108
  Not Assessed | 0 | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 37 | 34 | 33 | 17 | 121
  Puerto Rico | 1 | 3 | 5 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 6-Month Endpoint
Description: Values obtained from repeated measures analysis, which included the fixed categorical effects of treatment, baseline therapy strata (metformin versus diet and exercise [D&E]), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline glycosylated hemoglobin (HbA1c). Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 6 months
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline glycosylated hemoglobin (HbA1c) value.
Measure: Least Squares Mean (Standard Error); unit: percent glycosylated hemoglobin (HbA1c)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 24 | 21 | 23 | 12
percent glycosylated hemoglobin (HbA1c) | -0.08 (0.163) | 0.06 (0.179) | -0.15 (0.162) | 0.04 (0.234)
Statistical Analysis 1: Comparison: LY2428757 Plus TT223 3mg vs LY2428757 Plus TT223 Placebo; Test type: Superiority or Other; p = 0.623, Mixed Models Analysis — p-value is for LY2428757 plus TT223 3 mg versus LY2428757 plus TT223 placebo; Model included treatment, baseline therapy, strata, visit, and treatment-by-visit interaction, and continuous fixed covariate of baseline HbA1c
Statistical Analysis 2: Comparison: LY2428757 Plus TT223 2mg vs LY2428757 Plus TT223 Placebo; Test type: Superiority or Other; p = 0.809, Mixed Models Analysis — p-value is for LY2428757 plus TT223 2 mg versus LY2428757 plus TT223 placebo; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 4-Week Endpoint
Description: as for outcome 1
Time Frame: Baseline (Week -1), 4 weeks
Population: Intent-to-treat (ITT): All participants who received at least 1 dose of TT223 or its placebo with a baseline and at least 1 post-baseline glycosylated hemoglobin (HbA1c) value.
Measure: Least Squares Mean (Standard Error); unit: percent glycosylated hemoglobin (HbA1c)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 33 | 27 | 33 | 16
percent glycosylated hemoglobin (HbA1c) | -0.81 (0.111) | -0.97 (0.117) | -0.79 (0.112) | -0.19 (0.162)

3. Secondary Outcome: Change From Baseline in Mixed-Meal Tolerance Test (MMTT) Response - Glucose Area Under the Curve (AUC) at 3-Week and 6-Month Endpoints
Description: Standardized mixed-meal tolerance test (MMTT) used to assess changes in function of cells that make insulin (pancreatic beta cell function). Area under the plasma glucose concentration versus time curve calculated using linear-trapezoidal method. AUC for glucose represents area under curve of values when plotted over time. Larger area under the curve values represent greater average glucose value over time in response to meal. Least squares (LS) means adjusted for baseline, treatment, visit, treatment-by-visit. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 3 weeks, 6 months
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of TT223 or its placebo with both a baseline value and at least 1 post-baseline glucose area under the curve (AUC) value.
Measure: Least Squares Mean (Standard Error); unit: millimoles/liter*hour (mmol/L*hr)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 32 | 27 | 32 | 16
millimoles/liter*hour (mmol/L*hr)
  3 Weeks (n=32, 27, 32, 16) | 15.04 (2.121) | 13.14 (2.300) | 7.51 (2.138) | 28.47 (2.979)
  6 Months (n=23, 21, 22, 12) | -1.21 (1.490) | -1.05 (1.622) | -1.05 (1.549) | 1.46 (2.036)

4. Secondary Outcome: Change From Baseline in Mixed-Meal Tolerance Test (MMTT) Response - C-Peptide Area Under the Curve (AUC) at 3-Week and 6-Month Endpoints
Description: The area under the C-peptide concentration versus time curve was calculated using the linear-trapezoidal method. Area under the curve (AUC) for C-peptide represents area under the curve (AUC) of C-peptide values when plotted over time. Larger area under the curve (AUC) values represent a greater average C-peptide value over time in response to a meal. Least squares (LS) means adjusted for baseline, treatment, visit, treatment-by-visit interaction. Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 3 weeks, 6 months
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline C-peptide area under the curve (AUC) value.
Measure: Least Squares Mean (Standard Error); unit: millimoles/liter*hour (mmol/L*hr)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 32 | 28 | 32 | 16
millimoles/liter*hour (mmol/L*hr)
  3 Weeks (n=32, 28, 32, 16) | 44.44 (163.317) | -44.12 (176.487) | 119.23 (164.846) | -24.89 (226.274)
  6 Months (n=23, 21, 22, 12) | 221.02 (185.341) | -148.34 (197.247) | -241.88 (190.870) | -133.30 (253.264)

5. Secondary Outcome: Change From Baseline in Mixed Meal Tolerance Test (MMTT) Response - Ratio of Insulin Area Under the Curve (AUC)/Glucose Area Under the Curve (AUC) at 3-Week and 6-Month Endpoints
Description: Mixed meal tolerance test (MMTT) to assess changes in function of cells making insulin. AUCinsulin/AUCglucose ratio: index of insulin secretion. Larger values reflect greater secretion adjusted for glucose in response to meal. Area under insulin concentration versus time curve and area under plasma glucose concentration versus time curve calculated using linear-trapezoidal method. AUC for insulin and glucose represents AUC of values plotted over time. LS means adjusted for baseline, treatment, visit, treatment-by-visit. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 3 weeks, 6 months
Population: Intent-to-treat population (ITT): All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline AUC insulin/AUC glucose value. Reporting is on the 131 participants who received either TT223 or its placebo and reflects data only from the treatment and follow-up phases of the study.
Measure: Least Squares Mean (Standard Error); unit: millimoles/liter*hour (mmol/L*hr)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 30 | 27 | 32 | 16
millimoles/liter*hour (mmol/L*hr)
  3 Weeks (n=30, 27, 32, 16) | -0.96 (0.324) | -0.90 (0.341) | -0.16 (0.321) | -1.37 (0.433)
  6 Months (n=23, 21, 22, 12) | 0.05 (0.413) | -0.19 (0.425) | 0.15 (0.418) | -0.53 (0.566)

6. Secondary Outcome: Change From Baseline in Mixed-Meal Tolerance Test (MMTT) Response - Glucagon Area Under the Curve (AUC) at 3-Week and 6-Month Endpoints
Description: Standardized mixed meal tolerance test (MMTT) to assess changes in hormones in response to meal. Area under the plasma glucagon concentration versus time curve was calculated using the linear-trapezoidal method. Area under the curve (AUC) for glucagon represents the AUC of glucagon values when are plotted over time. Larger area under the curve (AUC) values represent a greater average glucagon value over time in response to a meal. Least squares (LS) means adjusted for baseline, treatment, visit, treatment-by-visit. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 3 weeks, 6 months
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of TT223 or its placebo with both a value at Week -1 and a value at that visit.
Measure: Least Squares Mean (Standard Error); unit: picomoles/liter (pmmol/L)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 30 | 28 | 32 | 16
picomoles/liter (pmmol/L)
  3 Weeks (n=30, 28, 32, 16) | -16.76 (15.367) | -29.12 (15.888) | -47.76 (14.890) | -26.46 (21.164)
  6 Months (n=23, 21, 22, 12) | -26.48 (4.504) | -15.96 (4.810) | -21.77 (4.654) | -12.10 (6.156)

7. Secondary Outcome: Change From Baseline in Mixed-Meal Tolerance Test (MMTT) Response - Glucagon-like Peptide-1 (GLP-1) Area Under the Cure (AUC) at 3-Week and 6-Month Endpoints
Description: Standardized mixed meal tolerance test (MMTT) to assess changes in hormones in response to meal. Area under plasma glucagon-like peptide-1 (GLP-1) concentration versus time curve calculated using linear-trapezoidal method. Area under the curve (AUC) for glucagon-like peptide-1 (GLP-1) represents the AUC of GLP-1 values when plotted over time. Larger AUC values represent a greater average GLP-1 value over time in response to meal. Least squares (LS) means adjusted for baseline, treatment, visit, treatment-by-visit. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 3 weeks, 6 months
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: picomoles/liter (pmmol/L)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 30 | 28 | 32 | 16
picomoles/liter (pmmol/L)
  3 Weeks (n=30, 28, 32, 16) | -0.90 (2.007) | 0.86 (2.094) | 1.48 (1.948) | -0.47 (2.702)
  6 Months (n=23, 21, 22, 12) | 0.41 (2.162) | 0.51 (2.302) | -5.93 (2.225) | 1.71 (2.955)

8. Secondary Outcome: Change From Baseline in Mixed-Meal Tolerance Test (MMTT) Response - Post-Prandial Glucose at 3-Week and 6-Month Endpoints
Description: Standardized MMTT to assess changes in function of cells that make insulin (pancreatic beta cells). Glucose measured at 2-hour timepoint during MMTT reflects glucose values in response to meal. Change in postprandial glucose calculated based on difference of 2-hour postprandial glucose at endpoint compared to baseline. Larger changes from baseline represent a greater postprandial glucose compared to 2-hour timepoint prior to treatment. Least squares (LS) means adjusted for baseline, treatment, visit, treatment-by-visit. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 3 weeks, 6 months
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of TT223 or its placebo with both a value at Week -1 and a value at that visit and time point being assessed.
Measure: Least Squares Mean (Standard Error); unit: millimoles/liter (mmol/L)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 32 | 27 | 31 | 16
millimoles/liter (mmol/L)
  3 Weeks 2 hours (n=32, 27, 31, 16) | -1.48 (0.417) | -1.12 (0.455) | -2.90 (0.426) | 0.60 (0.581)
  6 Months 2 hours (n=23, 21, 22, 12) | -0.72 (0.541) | -0.06 (0.576) | -0.43 (0.556) | 0.58 (0.748)

9. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at 4-Week and 6-Month Endpoints
Description: Values obtained from repeated measures analysis, which included the fixed categorical effects of treatment, baseline therapy strata (metformin versus diet and exercise [D&E]), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline fasting blood glucose (FBG). Fasting blood glucose (FBG) is the mixed meal tolerance test (MMTT) glucose assessment at time point 0, where available, otherwise it is the assessment taken from the chemistry panel. Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 4 weeks, 6 months
Population: Intent-to-treat (ITT): All participants who received at least 1 dose of TT223 or its placebo with a baseline and at least 1 post-baseline fasting blood glucose (FBG) value.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 32 | 27 | 33 | 16
millimoles per liter (mmol/L)
  4 weeks (n=32, 27, 33, 16) | -0.7 (0.40) | -1.6 (0.44) | -1.6 (0.40) | 0.5 (0.56)
  6 months (n=23, 21, 22, 12) | 0.1 (0.41) | 0.1 (0.44) | 0.3 (0.42) | -0.2 (0.57)

10. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1C) Adjusted for Baseline Glycosylated Hemoglobin (HbA1c), C-Peptide Level, Homeostasis Model Assessment of Insulin Resistance (HOMA), Duration of Diabetes, and Body Mass Index (BMI) at 6-Month Endpoint
Description: HbA1c adjusted: baseline HbA1c (<8%,≥8%); C-peptide level (normal, elevated); HOMA (<baseline median,≥baseline median); duration diabetes (<3,3-10,>10 years); BMI (<30,≥30). BMI estimates body fat based on weight/height squared. HOMA: index of function of cells that make insulin/insulin resistance. Indices derived from fasting glucose and insulin concentrations. LS means adjusted for treatment, baseline therapy, visit, treatment-by-visit, subgroup, subgroup-by-treatment, subgroup-by-visit, subgroup-by-treatment-by-visit. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 6 months
Population: Intent-to-treat (ITT): All participants who received at least 1 dose of TT223 or its placebo with a baseline and at least 1 post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: percent glucosylated hemoglobin (HbA1c)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 24 | 21 | 23 | 12
percent glucosylated hemoglobin (HbA1c)
  Baseline HbA1c <8% (n=24, 21, 23, 12) | -0.36 (0.169) | -0.22 (0.194) | -0.20 (0.183) | -0.53 (0.274)
  Baseline HbA1c >=8% (n=24, 21, 23, 12) | -0.17 (0.250) | 0.40 (0.228) | -0.12 (0.222) | 0.35 (0.269)
  C-peptide level normal (n=23, 21, 23, 12) | -0.26 (0.157) | 0.28 (0.165) | -0.20 (0.140) | -0.05 (0.195)
  C-peptide level elevated (n=23, 21, 23, 12) | -0.30 (0.254) | -0.78 (0.286) | 0.06 (0.600) | -0.32 (0.661)
  HOMA <baseline median (n=23, 19, 20, 12) | -0.18 (0.195) | 0.28 (0.241) | -0.23 (0.209) | 0.16 (0.227)
  HOMA >=baseline median (n=23, 19, 20, 12) | -0.24 (0.187) | -0.15 (0.188) | -0.38 (0.195) | -0.56 (0.322)
  BMI <30 (n=24, 21, 23, 12) | -0.45 (0.194) | 0.37 (0.250) | 0.07 (0.194) | -0.34 (0.335)
  BMI >=30 (n=24, 21, 23, 12) | -0.10 (0.179) | -0.12 (0.172) | -0.45 (0.189) | 0.03 (0.229)
  Duration of diabetes <3 years (n=24, 21, 23, 12) | -0.87 (0.348) | -0.77 (0.236) | 0.18 (0.240) | -0.49 (0.263)
  Duration diabetes 3-<10 years (n=24, 21, 23, 12) | -0.19 (0.157) | 0.50 (0.192) | -0.34 (0.172) | 0.49 (0.307)
  Duration of diabetes >=10 years (n=24, 21, 23, 12) | -0.19 (0.278) | 0.09 (0.349) | -0.50 (0.429) | -0.28 (0.425)

11. Secondary Outcome: Change From Baseline in MMTT Response (Postprandial Glucose, Glucose AUC, Insulin/c-Peptide Secretory Response, HOMA, GLP-1, Glucagon) Adjusted for Baseline HbA1c, C-Peptide Level, HOMA, Duration of Diabetes, Weight at Week 0, 3, Month 3.5, 6 Endpoints
Description: Subgroup analyses for mixed meal tolerance test (MMTT) response (adjusted for baseline glycosylated hemoglobin (HbA1c), C-peptide level, Homeostasis Model Assessment of Insulin Resistance (HOMA), duration of diabetes, weight) not performed due to lack of statistically significant findings in subgroup analysis for HbA1c analyses. HOMA was not done for mixed meal tolerance test (MMTT) because it is not calculated from the mixed meal tolerance test (MMTT). It is reported separately as a secondary outcome measure. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), Week 0, 3 weeks, 3.5 months, 6 months
Population: Because the subgroup analyses for MMTT response were not conducted due to the lack of statistically significant findings in the subgroup analysis for the HbA1c analyses, zero participants were analyzed.
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) Adjusted for Baseline HbA1c, C-Peptide Level, Homeostasis Model Assessment of Insulin Resistance, Duration of Diabetes, and Weight at 3-Week, 4-Week, 2-Month, 3.5-Month, 5-Month, and 6-Month Endpoints
Description: The subgroup analyses for fasting blood glucose (FBG) (adjusted for baseline glycosylated hemoglobin [HbA1c]), C-peptide level, homeostasis model assessment of insulin resistance (HOMA), duration of diabetes, and weight) were not performed due to the lack of statistically significant findings in the subgroup analysis for the glycosylated hemoglobin (HbA1c) analyses. Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 3 weeks, 4 weeks, 2 months, 3.5 months, 5 months, 6 months
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Mean Change From Baseline in Weight at Week 0, Week 4, and 6-Month Endpoints
Description: Values obtained from repeated measures analysis, which included the fixed categorical effects of treatment, baseline therapy strata (metformin versus diet and exercise [D&E]), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline weight. Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), Week 0, 4 weeks, 6 months
Population: Intent-to-treat (ITT): All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline weight value.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 38 | 37 | 38 | 18
kilograms (kg)
  Week 0 (n=38, 37, 38, 18) | -0.198 (0.2380) | -0.137 (0.2455) | -0.288 (0.2438) | 0.305 (0.3338)
  4 weeks (n=33, 27, 33, 16) | -0.561 (0.2923) | -0.975 (0.3167) | -0.824 (0.2956) | -0.542 (0.4090)
  6 months (n=24, 21, 23,12) | 0.066 (0.7007) | 0.026 (0.7613) | -0.762 (0.7044) | -0.164 (0.9996)

14. Secondary Outcome: Number of Participants With Antibodies to LY2428757
Description: Participants who were positive for antibodies to LY2428757.
Time Frame: Baseline (Week -1) through 6 months
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline value.
Measure: Number; unit: participants
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 38 | 37 | 38 | 18
participants | 1 | 1 | 0 | 0

15. Secondary Outcome: Number of Participants With Antibodies to TT223
Description: Participants who were positive for antibodies for TT223.
Time Frame: Baseline (Week -1) through 6 months
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 38 | 37 | 38 | 18
participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Pharmacokinetics (PKs) of TT223, First Dose - Time of Maximum Observed Drug Concentration (Tmax)
Description: Time of maximum observed drug concentration (Tmax) is the time at which the maximum observed concentration (Cmax) occurs.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: hours
Groups:
- LY2428757 Plus TT223 2 mg: Weekly LY2428757 14 mg subcutaneous injection for 5 weeks plus TT223 2 mg subcutaneous injection daily for 4 weeks
- LY2428757 Plus TT223 3 mg: Weekly LY2428757 14 mg subcutaneous injection for 5 weeks plus TT223 3 mg subcutaneous injection daily for 4 weeks
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 35 | 33
hours | 0.50 (0.30-3.00) [0.30 to 3.00] | 1.00 (0.30-4.00) [0.30 to 4.00]

17. Secondary Outcome: Pharmacokinetics (PKs) of TT223, First Dose - Maximum Observed Drug Concentration (Cmax)
Description: Maximum observed drug concentration (Cmax) is the maximum observed concentration of drug.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/ml)
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 35 | 33
nanograms per milliliter (ng/ml) | 8.52 (276) | 8.46 (531)

18. Secondary Outcome: Pharmacokinetics (PKs) of TT223, First Dose - Half-Life (t1/2) Associated With the Terminal Rate Constant (λz) in Non-Compartmental Analysis
Description: Half-life is the time it takes for the concentration of drug in plasma to decline by 50%.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 35 | 33
hours | 1.11 (56) | 1.20 (70)

19. Secondary Outcome: Pharmacokinetics (PKs) of TT223, First Dose - Area Under the Curve (AUC)(0-infinity)
Description: Area under the curve (AUC)(0-infinity) = area under concentration versus time from zero to infinity. Area under the curve (AUC) is a measure of the total exposure to a drug.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/ml)
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 35 | 33
nanograms*hour/milliliter (ng*hr/ml) | 28.0 (66) | 52.2 (38)

20. Secondary Outcome: Pharmacokinetics (PKs) of TT223, First Dose - Apparent Total Body Clearance of Drug Calculated After Extra-Vascular Administration (CL/F)
Description: Apparent total body clearance of drug calculated after extra-Vascular administration (CL/F) is the apparent volume of the body fluid cleared of the drug per unit of time, adjusted for how much drug goes into the body fluid.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour (L/hr)
Groups:
- LY2428757 Plus TT223 3 mg: Weekly LY2428757 14 mg subcutaneous injection for 5 weeks plus TT223 3 mg subcutaneous injection daily for 4 weeks TT223
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 35 | 33
liters/hour (L/hr) | 71.4 (66) | 57.5 (38)

21. Secondary Outcome: Pharmacokinetics (PKs) of TT223, First Dose - Apparent Volume of Distribution During the Terminal Phase After Extra-Vascular Administration (Vz/F), Apparent Volume of Distribution at Steady-State After Extra-Vascular Administration (Vss/F)
Description: volume of distribution during the terminal phase after extra-vascular administration (Vz/F): Apparent volume that contains drug after absorption is complete and drug is no longer being given. Apparent volume of distribution at steady-State after extra-vascular administration (Vss/F): Apparent volume that contains drug when drug is being given continuously.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 35 | 33
liters (L)
  Vz/F | 115 (108) | 99.2 (87)
  Vss/F | 157 (91) | 136 (60)

22. Secondary Outcome: Pharmacokinetics (PKs) of TT223, 3-Week Time Point - Maximum Observed Drug Concentration (Cmax)
Description: Maximum observed drug concentration (Cmax) is the maximum observed concentration of drug.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/ml)
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 26 | 25
nanograms per milliliter (ng/ml) | 5.61 (652) | 5.97 (1320)

23. Secondary Outcome: Pharmacokinetics (PKs) of TT223, 3-Week Time Point - Time of Maximum Observed Drug Concentration (Tmax)
Description: as for outcome 16
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 26 | 25
hours | 0.50 [0.33 to 6.00] | 0.50 [0.32 to 6.00]

24. Secondary Outcome: Pharmacokinetics (PKs) of TT223, 3-Week Time Point - Half Life (t1/2)
Description: Half-life (t1/2) is the time it takes for the concentration of drug in plasma to decline by 50%.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 26 | 25
hours | 1.08 (59) | 1.03 (52)

25. Secondary Outcome: Pharmacokinetics (PKs) of TT223, 3-Week Time Point - Area Under Concentration Versus Time From Zero to Infinity (AUC[0-infinity])
Description: Area under concentration versus time curve from zero to infinity (AUC[0-infinity]). Area under the curve (AUC) is a measure of the total exposure to a drug.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*hr/ml)
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 26 | 25
nanograms*hour/milliliter (ng*hr/ml) | 25.1 (67) | 32.6 (596)

26. Secondary Outcome: Pharmacokinetics (PKs) of TT223, 3-Week Time Point - Apparent Total Body Clearance of Drug Calculated After Extra-Vascular Administration (CL/F)
Description: as for outcome 20
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 26 | 25
liters per hour (L/hr) | 79.6 (67) | 92.3 (596)

27. Secondary Outcome: Pharmacokinetics (PKs) of TT223, 3-Week Time Point - Apparent Volume of Distribution During the Terminal Phase After Extra-Vascular Administration (Vz/F), Apparent Volume of Distribution at Steady-State After Extra-Vascular Administration (Vss/F)
Description: Apparent volume of distribution during the terminal phase after extra-vascular administration (Vz/F) is the apparent volume that contains drug after absorption is complete and drug is no longer being given. Apparent volume of distribution at steady-state after extra-vascular administration (Vss/F) is the apparent volume that contains drug when drug is being given continuously.
Time Frame: 0 (pre-dose), 0.33, 0.5, 1, 2, 3, 4, 6 hours
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | LY2428757 Plus TT223 2 mg | LY2428757 Plus TT223 3 mg
Number analyzed (Participants) | 26 | 25
liters (L)
  Vz/F | 124 (129) | 137 (645)
  Vss/F | 163 (97) | 202 (519)

28. Secondary Outcome: Pharmacokinetics (PKs) of LY2428757, 3-Week Time Point - Maximum Observed Drug Concentration (Cmax)
Description: Maximum observed drug concentration (Cmax) is the maximum observed concentration of drug. LY2428757 concentrations were collected at only a single timepoint; therefore, pharmacokinetic (PK) parameters could not be modeled from the data. Analysis was not done due to insufficient time points being collected.
Time Frame: 0 (pre-dose)
Population: Analyses were not conducted due to insufficient time points being collected; zero participants were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/ml)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

29. Secondary Outcome: Visual Analog Scale (VAS) for Nausea
Description: The Visual Analog Scale (VAS) is a continuous measure for degree of nausea and/or gastrointestinal discomfort. Each of these scales is 100 millimeters (mm) in length with 0 meaning no nausea at all and 100 meaning extreme nausea. Participants record self-assessment of how much nausea they have had, from 0 to 100, during the time interval indicated.
Time Frame: 4 weeks, 6 months
Population: Each visit includes participants who received at least 1 dose of TT223 or its placebo who had both a baseline value and a value at that visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 38 | 37 | 38 | 18
units on a scale
  Baseline (n=38, 37, 38, 18) | 10.8 (19.21) | 5.7 (11.27) | 8.4 (17.12) | 4.7 (11.15)
  4 weeks (n=33, 27, 34, 16) | 22.0 (20.49) | 27.6 (26.67) | 11.9 (19.66) | 9.1 (11.92)
  6 months (n=27, 24, 30, 15) | 7.1 (11.31) | 3.4 (4.86) | 7.3 (18.38) | 8.1 (12.99)

30. Secondary Outcome: Change From Baseline in Waist Circumference at 6-Month Endpoint
Description: Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 6 months
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 31 | 35 | 28 | 13
centimeters (cm) | 1.55 (5.276) | -0.60 (2.433) | -0.16 (2.599) | -0.33 (3.060)

31. Secondary Outcome: 7-point Profile, Self-Monitored Blood Glucose (SMBG) Values
Description: The 7-point average is the average of the mean value of all time points for the visit. Time points included pre-morning meal, 2 hours after morning meal, pre-midday meal, 2 hours after midday meal, pre-evening meal, 2 hours after evening meal, and bedtime.
Time Frame: Baseline (Week -1), 4 weeks, 6 months
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 31 | 22 | 30 | 15
milligrams per deciliter (mg/dL)
  4 weeks (n=31, 22, 30, 15) | 152.75 (29.973) | 147.10 (24.514) | 142.38 (32.199) | 169.23 (55.866)
  6 months (n=24, 19, 23, 12) | 173.18 (46.455) | 177.50 (49.379) | 176.33 (38.900) | 172.05 (28.688)

32. Secondary Outcome: Change From Baseline in 7-Point Profile, Self-Monitored Blood Glucose (SMBG) at 4-Week and 6-Month Endpoints
Description: 7-point average=average of mean value of all time points for visit (premorning meal, 2-hours postmorning meal, premidday meal, 2-hours postmidday meal, preevening meal, 2-hours postevening meal, bedtime). Values represent mean of values collected same time on 3 separate days within week prior to visit. Values from repeated measures included fixed categorical effects: treatment, baseline therapy strata, visit, treatment-by-visit, continuous fixed covariate baseline <7-point average glucose value or time point presented. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 4 weeks, 6 months
Population: Intent-to-treat (ITT): All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline value for the variable being analyzed.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 31 | 22 | 30 | 15
milligrams per deciliter (mg/dL)
  Average 4 weeks (n=31,22,30,15) | -29.28 (5.082) | -45.03 (6.192) | -41.18 (5.215) | -18.95 (7.136)
  Pre-morning meal fasting 4 weeks (n=31,22,30,15) | -24.30 (5.335) | -42.95 (6.526) | -32.41 (5.466) | -5.89 (7.529)
  2 hours after morning meal 4 weeks (n=30,21,29,15) | -38.41 (6.094) | -63.72 (7.409) | -51.70 (6.158) | -23.80 (8.313)
  Pre-midday meal 4 weeks (n=30,22,29,15) | -14.76 (5.950) | -30.83 (7.088) | -32.86 (6.048) | -14.96 (8.194)
  2 hours after midday meal 4 weeks (n=30,22,29,15) | -32.64 (6.719) | -38.90 (8.037) | -39.30 (6.907) | -22.19 (9.328)
  Pre-evening meal 4 weeks (n=30,22,29,15) | -26.67 (5.565) | -28.36 (6.663) | -30.87 (5.760) | -16.85 (7.721)
  2 hours after evening meal 4 weeks (n=30,22,29,14) | -37.72 (6.728) | -53.39 (8.125) | -51.07 (6.927) | -29.01 (9.574)
  Bedtime 4 weeks (n=28,21,28,15) | -35.44 (7.112) | -44.50 (8.378) | -41.22 (7.108) | -14.66 (9.492)
  Average 6 months (n=24,19,23,12) | -7.66 (7.693) | -11.70 (8.759) | -5.76 (7.970) | -13.07 (10.751)
  Pre-morning meal fasting 6 months (n=24,19,23,12) | -5.00 (5.981) | -4.89 (6.869) | -10.48 (6.236) | -6.45 (8.314)
  2hours after morning meal 6 months (n=23,19,23,12) | -12.25 (8.654) | -18.40 (9.631) | -14.84 (8.739) | -27.48 (11.755)
  Pre-midday meal 6 months (n=24,19,23,12) | -4.76 (8.345) | 3.95 (9.452) | -0.96 (8.558) | -9.54 (11.554)
  2hours after midday meal 6 months (n=24,19,23,12) | -5.51 (9.418) | -4.15 (10.722) | 4.67 (9.788) | -12.71 (13.152)
  Pre-evening meal 6 months (n=24,19,23,12) | -2.61 (8.562) | -7.53 (9.727) | 1.53 (8.881) | -15.57 (11.958)
  2hours after evening meal 6 months (n=24,19,23,12) | -11.20 (10.373) | -20.89 (11.815) | -9.98 (10.726) | -7.62 (14.491)
  Bedtime 6 months (n=21,18,22,11) | -11.27 (9.684) | -21.61 (10.612) | -6.40 (9.599) | -3.79 (13.150)

33. Secondary Outcome: Change From Baseline in Lipase at Week 0, Week 4, and 6-Month Endpoints
Description: Values obtained from repeated measures analysis, which included the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline serum lipase. Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), Week 0, 4 weeks, 6 months
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: units per liter (U/L)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 38 | 36 | 38 | 18
units per liter (U/L)
  Week 0 (n=38, 36, 38, 18) | 12.1 (7.89) | 8.1 (8.11) | 15.8 (7.89) | 2.3 (11.46)
  4 weeks (n=32, 27, 34, 16) | 14.8 (9.92) | 10.1 (10.53) | 40.5 (9.79) | 0.4 (14.24)
  6 months (n=28, 23, 30, 15) | -2.1 (4.52) | -5.0 (4.95) | 7.0 (4.42) | -3.1 (6.34)

34. Secondary Outcome: Change From Baseline in Amylase at 6-Month Endpoint
Description: Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 6 months
Population: Intent-to-treat (ITT): All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline amylase value.
Measure: Least Squares Mean (Standard Error); unit: units/liter (U/L)
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 27 | 23 | 30 | 15
units/liter (U/L) | -2.9 (3.15) | -4.5 (3.45) | 1.5 (3.01) | -10.3 (4.23)

35. Secondary Outcome: Percentage of Participants With 2-Fold Elevation of Lipase and/or Amylase at Any Timepoint
Description: Values obtained from repeated measures analysis, which included the fixed categorical effects of treatment, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline amylase.
Time Frame: Baseline (Week -1) through 6 months
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 38 | 37 | 38 | 18
percentage of participants
  Lipase >= 2 times the upper limit of normal | 0 | 0 | 2 | 0
  Amylase >=2 times the upper limit of normal | 0 | 0 | 0 | 0

36. Secondary Outcome: Percentage of Participants With Hypoglycemia
Description: Calculation of frequency of low glucose for time period. Hypoglycemia≥1 events: severe<50mg/dL, unable to treat self/recover after treatment; documented symptomatic≤70mg/dL, adrenergic/neuroglycopenic symptoms; asymptomatic≤70mg/dL no symptoms; probable symptomatic glucose missing, adrenergic/neuroglycopenic symptoms; relative>70mg/dL, adrenergic/neuroglycopenic symptoms, nocturnal≤70mg/dL, adrenergic/neuroglycopenic symptoms between bedtime/waking. Because number participants who experienced hypoglycemia was low for every arm (1-3/arm) did not model percentage participants with hypoglycemia.
Time Frame: Baseline (Week -1) through 6 months
Population: Because the number of hypoglycemia events were too low to model the percentage of hypoglycemia, zero participants were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

37. Secondary Outcome: Number of Participants With Hypoglycemia
Description: The number of participants for whom low blood glucose was reported. Hypoglycemia ≥1 events including: severe hypoglycemia(glucose <50mg/dL, unable to treat self or recover after treatment); documented symptomatic (glucose ≤70mg/dL, adrenergic or neuroglycopenic symptoms); asymptomatic (glucose ≤70mg/dL no symptoms); probable symptomatic (glucose missing, adrenergic or neuroglycopenic symptoms); relative (glucose >70mg/dL, adrenergic or neuroglycopenic symptoms), nocturnal (glucose ≤70mg/dL, adrenergic or neuroglycopenic symptoms between bedtime/waking).
Time Frame: Baseline (Week -1) through 6 months
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 38 | 37 | 38 | 18
participants | 2 | 2 | 3 | 1

38. Secondary Outcome: Number of Participants With Adjudicated and Confirmed Deaths and Non-Fatal Cardiovascular (CV) Events at Any Timepoint
Description: The protocol specified that deaths and nonfatal cardiovascular (CV) adverse events (AEs) be adjudicated by independent physician(s) with cardiology or neurology experience. The CV AEs to be adjudicated were protocol-defined as myocardial infarction (MI), hospitalization for unstable angina or for heart failure, coronary interventions (coronary artery bypass graft or percutaneous coronary intervention [PCI]) and cerebrovascular events including cerebrovascular accident (stroke) and transient ischemic attack (TIA). 3 CV events were adjudicated by an external independent adjudication committee.
Time Frame: Baseline (Week -1) through 6 months
Population: All participants who received at least 1 dose of TT223 or its placebo.
Measure: Number; unit: participants
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 38 | 37 | 38 | 18
participants | 2 | 0 | 0 | 1

39. Secondary Outcome: Change From Baseline in Fasting Insulin at 4-Week and 6-Month Endpoints
Description: Values obtained from repeated measures analysis, which included the fixed categorical effects of treatment, baseline therapy strata (metformin versus diet and exercise [D&E]), visit, and treatment-by-visit interaction, as well as the continuous, fixed covariate of baseline Fasting Insulin. Fasting insulin is the Mixed-Meal Tolerance Test (MMTT) insulin assessment at timepoint 0, where available, otherwise it is the assessment taken from the fasting laboratory measurements obtained during the clinic visit. Change from baseline means the absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 4 weeks, 6 months
Population: Intent-to-treat: All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline fasting insulin value.
Measure: Least Squares Mean (Standard Error); unit: microinternational units/milliliter
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 31 | 25 | 32 | 16
microinternational units/milliliter
  4 weeks (n=31, 25, 32, 16) | 6.7 (4.57) | -4.2 (4.89) | 4.7 (4.49) | 0.7 (6.21)
  6 months (n=23, 20, 22, 12) | 2.3 (4.03) | -4.2 (4.41) | 2.8 (3.95) | -7.2 (5.43)

40. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment (HOMA) at 3-Week and 6-Month Endpoints
Description: Values from repeated measures include fixed categorical effects of treatment, baseline therapy strata, visit, treatment-by-visit, continuous fixed covariate of baseline HOMA derived beta-cell function (HOMA-B). HOMA=index of function of cells that make insulin. Indices derived from fasting glucose and insulin concentrations. HOMA is measurement reflecting fasting plasma glucose and insulin. Has no defined minimum/maximum value. HOMA-B values generated from table reflecting values derived from Oxford HOMA2 model calculator. Change from baseline=absolute change from baseline (endpoint-baseline).
Time Frame: Baseline (Week -1), 3 weeks, 6 months
Population: Intent-to-treat: All participants who received at least 1 dose of TT223 or its placebo with both a baseline and at least 1 post-baseline HOMA value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Number analyzed (Participants) | 26 | 23 | 26 | 14
units on a scale
  3 weeks (n=26, 23, 26, 14) | 19.12 (7.605) | 34.73 (8.093) | 37.76 (7.597) | -14.99 (10.193)
  6 months (n=19, 18, 19, 11) | -3.05 (9.128) | 4.41 (9.415) | 19.17 (9.111) | -9.01 (11.986)

ADVERSE EVENTS:
Arm/Group | LY2428757 Plus TT223 3mg | LY2428757 Plus TT223 2mg | LY2428757 Plus TT223 Placebo | LY Placebo Plus TT223 Placebo
Serious Adverse Events (participants affected / at risk) | 2/38 | 1/37 | 0/38 | 2/18
Other Adverse Events (participants affected / at risk) | 23/38 | 29/37 | 26/38 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2428757 Plus TT223 3mg (N=38) | LY2428757 Plus TT223 2mg (N=37) | LY2428757 Plus TT223 Placebo (N=38) | LY Placebo Plus TT223 Placebo (N=18)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2428757 Plus TT223 3mg (N=38) | LY2428757 Plus TT223 2mg (N=37) | LY2428757 Plus TT223 Placebo (N=38) | LY Placebo Plus TT223 Placebo (N=18)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (14) | 15 (22) | 5 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 5 (11) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days